CLINICAL TRIAL: NCT04510558
Title: Reducing the Incidence of Incisional Hernia After Stoma Closure Using a PROphylactic MESH: a Single-blinded Randomized Controlled Trial (PROMESH TRIAL).
Brief Title: Reducing the Incidence of Incisional Hernia After Stoma Closure Using a Prophylactic Mesh
Acronym: PROMESH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jeremy Meyer, Consultant surgeon, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROMESH TRIAL
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Incisional Hernia
Keywords: mesh; ileostomy; colostomy; stoma closure
MeSH Terms: conditions — Incisional Hernia | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Intervention Model Description: Patients will be recruited during the preoperative consultation. Patients will be given written information related to the study and will sign an informed consent form. Investigators will be contacted and perform randomization using the RedCap (Research Electronic Data Capture) software system on a 1:1 allocation ratio between study groups. The surgery planning form will be forwarded to the investigators, which will indicate if a mesh should be added or not to the stoma closure procedure.
Who Masked: Participant
Masking Description: Patients will be blinded for the study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (mesh) (Experimental): Insertion of a non-resorbable mesh in the subway position.
  Interventions: Device: Stoma closure with non-resorbable mesh (ULTRAPRO Advanced Mesh, Ethicon, Johnson & Johnson) in the sublay position
- Control (no mesh) (Sham Comparator): No insertion of mesh.
  Interventions: Procedure: Stoma closure without mesh

INTERVENTIONS:
Device: Stoma closure with non-resorbable mesh (ULTRAPRO Advanced Mesh, Ethicon, Johnson & Johnson) in the sublay position — * Antibioprophylaxis using cefuroxime and metronidazole
  * Standard disinfection and sterile draping
  * Circular incision around the stoma using the scalpel blade
  * Dissection around the stoma until entering the abdominal cavity
  * Closure of the stoma using a linear stapler
  * A midline laparotomy may be performed or not
  * Realization of an extra-corporeal or intra-corporeal side-to-side handsewn anastomosis
  * Closure of the posterior aponeurosis using separate Maxon 2-0 stitches
  * Application of an ULTRAPRO Advanced Mesh, Ethicon, Johnson & Johnson, with +2cm on the edges, secured by 4 stiches of Maxon 2-0
  * Closure of the anterior aponeurosis using separate Maxon 2-0 stitches
  * No subcutaneous stitches
  * Partial purse string skin closure using Monocryl 3-0
  * Standard wound dressing
  Arms: Intervention (mesh)
Procedure: Stoma closure without mesh — * Antibioprophylaxis using cefuroxime and metronidazole
  * Standard disinfection and sterile draping
  * Circular incision around the stoma using the scalpel blade
  * Dissection around the stoma until entering the abdominal cavity
  * Closure of the stoma using a linear stapler
  * A midline laparotomy may be performed or not
  * Realization of an extra-corporeal or intra-corporeal side-to-side handsewn anastomosis
  * Closure of the posterior aponeurosis using separate Maxon 2-0 stitches
  * Closure of the anterior aponeurosis using separate Maxon 2-0 stitches
  * No subcutaneous stitches
  * Partial purse string skin closure using Monocryl 3-0
  * Standard wound dressing
  Arms: Control (no mesh)

SUMMARY:
Background:

Preliminary studies have shown that application of a prophylactic mesh during stoma closure reduces the incidence of incisional hernia at site of stoma closure.

Methods/Design:

The study will be a randomized controlled single-blinded monocentric study determining the 1-year incidence of incisional hernia in cancer patients undergoing ileostomy or colostomy closure with or without prophylactic non-absorbable mesh applied in the sublay position.

Discussion:

Prevention of incisional hernia at site of stoma closure will lead to an improvement in patients' quality of life and generating savings for healthcare systems. To date, no randomized controlled trial assessing the effect of prophylactic mesh applied during stoma closure on the prevention of incisional hernia has been published. With the present randomized controlled trial, we expect to demonstrate that the application of a prophylactic mesh reduces the one-year incidence of incisional hernia at site of stoma closure.

DETAILED DESCRIPTION:
Background:

Recent pooled evidence indicates that the incidence of incisional hernia after stoma closure is of 7.4%, but this finding is limited by an important heterogeneity (reported incidences ranging from 0 to 48%). The pooled incidence of incisional hernia ranges from 4 to 10% according to the type of stoma, with the highest incidence reported after colostomy closure (10%). These incisional hernias at site of stoma generate patient discomfort, alteration of quality of life, complications such as bowel occlusion and increased costs for healthcare systems.

Several retrospective studies have investigated the impact of a prophylactic mesh during stoma closure on the incidence of incisional hernia. For instance, Liu et al. compared 47 patients who benefited from ileostomy closure with a synthetic non-resorbable mesh with 36 patients who underwent the same surgery without mesh, and found that incidences of incisional hernia (with a median follow-up of 18 months) were of 6.4% and 36.1%, respectively 3. Similarly, a retrospective case-control study compared 30 patients who had ileostomy closure with prophylactic biological mesh with 30 matched patients without mesh. At one year, the incidence of incisional hernia diagnosed with CTscan was of 3.3% in patients with mesh versus 40% in patients without mesh 4. A multicenter randomized controlled trial (RCT) is currently underway to evaluate whether an intra-abdominal mesh allows to prevent the one year incidence of CTscan-proven incisional hernia in patients undergoing ileostomy and colostomy closures 5. A preliminary feasibility study demonstrated the safety of the procedure 6. However, no specific techniques for mesh fixation and position are documented in the RCT protocol, which might introduce confusion factors in the final analysis. Further, applying an intra-abdominal mesh might potentially result in long-term complications due to bowel adhesion to the abdominal wall.

Therefore, we have planned to undertake a RCT aiming at determining whether a prophylactic non-resorbable mesh in the sublay position allows or not reducing the incidence of incisional hernia after ileostomy or colostomy closure.

Methods/Design:

Study design:

The study will be a randomized controlled single-blinded monocentric study determining the one year incidence of incisional hernia in patients undergoing ileostomy or colostomy closure with or without prophylactic mesh.

Study setting:

The study will take place at the Division of Digestive Surgery, University Hospitals of Geneva, Geneva, Switzerland.

Population:

Adult patients undergoing ileostomy or colostomy closure after surgery for digestive cancer will be considered as eligible for the study.

Inclusion criteria:

* Adult patient
* Ileostomy or colostomy performed during surgery for digestive cancer
* Planned elective closure of ileostomy or colostomy
* Informed written consent

Exclusion criteria:

* Allergy to mesh
* Patients under corticosteroids or other immunosuppressive treatment
* Inability/refusal to follow the procedures of the study

Drop-outs:

* Stoma closure not performed
* One-year follow-up not completed
* Withdrawal of consent
* Redo surgery at the site of stoma not related to the mesh and/or to incisional hernia
* Violation of protocol

Intervention: Stoma closure with non-resorbable mesh in the sublay position

* Antibioprophylaxis using cefuroxime and metronidazole
* Standard disinfection and sterile draping
* Circular incision around the stoma using the scalpel blade
* Dissection around the stoma until entering the abdominal cavity
* Closure of the stoma using a linear stapler
* A midline laparotomy may be performed or not
* Realization of an extra-corporeal or intra-corporeal side-to-side handsewn anastomosis
* Closure of the posterior aponeurosis using separate Maxon 2-0 stitches
* Application of an ULTRAPRO Advanced Mesh, Ethicon, Johnson & Johnson, with +2cm on the edges, secured by 4 stiches of Maxon 2-0
* Closure of the anterior aponeurosis using separate Maxon 2-0 stitches
* No subcutaneous stitches
* Partial purse string skin closure using Monocryl 3-0
* Standard wound dressing

Control: Stoma closure without mesh

* Antibioprophylaxis using cefuroxime and metronidazole
* Standard disinfection and sterile draping
* Circular incision around the stoma using the scalpel blade
* Dissection around the stoma until entering the abdominal cavity
* Closure of the stoma using a linear stapler
* A midline laparotomy may be performed or not
* Realization of an extra-corporeal or intra-corporeal side-to-side handsewn anastomosis
* Closure of the posterior aponeurosis using separate Maxon 2-0 stitches
* Closure of the anterior aponeurosis using separate Maxon 2-0 stitches
* No subcutaneous stitches
* Partial purse string skin closure using Monocryl 3-0
* Standard wound dressing

Outcomes:

Primary outcome:

The primary outcome will be the incidence of incisional hernia at site of stoma at one year after closure. The presence or not of an incisional hernia will be assessed clinically by a specialist in general surgery and radiologically by computed tomography realized in the setting of cancer follow-up. The investigator performing the one-year follow-up and the radiologist interpreting the CTscan will be blinded for the study group. Patients diagnosed with incisional hernia and/or reoperated for a complication related to stoma closure and/or mesh will be considered as treatment failure.

Secondary outcome:

The secondary outcome will be the incidence of surgical site infection (SSI) at site of stoma closure, evaluated at 7 and at 31 days after stoma closure according to the Center for Disease Control definition. Specialized nurses will record pictures of the stoma site for blinded evaluation by an investigator. In case of occurrence, SSI will be treated according to institutional guidelines.

Randomization, allocation concealment and blinding :

Patients will be recruited during the preoperative consultation. Patients will be given written information related to the study and will sign an informed consent form. Investigators will be contacted and perform randomization using the RedCap (Research Electronic Data Capture) software system on a 1:1 allocation ratio between study groups. The surgery planning form will be forwarded to the investigators, which will indicate if a mesh should be added or not to the stoma closure procedure. Patients will be blinded for the study group.

Sample size calculation:

Considering the results of existing studies comparing the incidence of incisional hernia after stoma closure with and without prophylactic mesh, we aimed reducing the incidence of incisional hernia from 30% to 5%. Using the two-sided Pearson's chi-squared test for proportions, with a power set at 0.8 and an alpha at 0.05, and considering a 1:1 allocation ratio, we will have to include 72 patients (36 with mesh and 36 without mesh).

Variables of interest:

Variables of interest will be recorded by the investigator into a case-report form generated in the RedCap software.

Variables related to stoma confection:

* Date of stoma confection
* Age
* Gender
* BMI
* ASA class
* Tobacco use
* Pre-albumin concentration
* Albumin concentration
* Proteins concentration
* Neo-adjuvant treatment
* Surgery performed in emergency or elective setting
* Diagnostic
* Type of surgery performed
* Type of stoma
* Site of stoma
* Length of stay

Variables related to stoma closure:

* Date of stoma closure
* Age
* BMI
* ASA class
* Tobacco use
* Pre-albumin concentration
* Albumin concentration
* Proteins concentration
* Type of surgery performed
* Presence or not of a parastomal hernia
* Length of stay

Variables related to follow-up at 7 days after the stoma closure:

* Date of early follow-up
* Presence or not of a SSI
* Pictures of the stoma site

Variables related to follow-up at 1 year after stoma closure:

* Date of late follow-up
* Age
* BMI
* Adjuvant treatment
* Presence or not of an incisional hernia at the site of stoma closure (clinical examination)
* Presence or not of an incisional hernia at the site of stoma closure (CTscan)
* If appropriate, variables related to the management of the incisional hernia

Statistical analysis :

Continuous variables will be expressed as medians±SD. Categorical variables will be expressed as numbers (proportions). Continuous variables and outcomes will be compared using the two-sided Student's t test. Categorical variables and outcomes will be compared using the Chi-square test or the exact Fisher test, when appropriate. Subgroup analyses will be performed according to BMI class and type of stoma. An in interim analysis will be performed when 36 patients are included; if a difference >15% of SSI (the short-term outcome) between the 2 groups is put observed, the study will be terminated. A p-value <0.05 will be considered as significant. Analyses will be performed using GraphPad Prism version 15 and STATA version 13.

Discussion:

Existing literature reports heterogeneous incidences of incisional hernia at stoma site after stoma closure. Several systematic reviews and meta-analyses, however, documented clinically significant pooled incidences 1, 2. Considering that the incisional hernia usually requires surgery and hospitalization, we believe that this complication, in addition to altering patients' quality of life, also impairs healthcare systems budgets.

Preliminary studies have shown that insertion of a prophylactic mesh, resorbable or not, during stoma closure, reduces the incidence of incisional hernia at stoma site 3, 4. However, to date, no RCT has been released on the subject. Further, the procedure seems to be safe, with very few SSI reported.

The aim of the present RCT will be to determine whether application of a prophylactic non-absorbable mesh during stoma closure allows or not for the prevention of incisional hernia at one year. Subgroup analysis will be performed according to the type of stoma and to BMI class. Furthermore, secondary analysis of the results might allow us to gather enough data for an objective cost-benefit analysis of the technique.

The strengths of the present RCT will be the following : (1) Good external validity due to the representation of all types of stomas, (2) Mesh in the sublay position, where the risk of intra-abdominal complications is lower and application is the easiest (as compared to intra-abdominal mesh), (3) Use of an affordable mesh (as compared to biological mesh), (5) assessment of the presence or not of incisional hernia by CTscan.

Trial status:

The RCT protocol was accepted by the local ethical committee.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Ileostomy or colostomy performed during surgery for digestive cancer
* Planned elective closure of ileostomy or colostomy
* Informed written consent

Exclusion Criteria:

* Allergy to the mesh
* Patients under corticosteroids or other immunosuppressive treatment
* Inability/refusal to follow the procedures of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of incisional hernia at site of stoma at one year after closure | At one year after stoma closure
  The presence or not of an incisional hernia will be assessed clinically by a specialist in general surgery and radiologically by computed tomography realized in the setting of cancer followup. The investigator performing the 1-year follow-up and the radiologist interpreting the CTscan will be blinded for the study group. Patients diagnosed with incisional hernia and/or reoperated for a complication related to stoma closure and/or mesh will be considered as treatment failure.

SECONDARY OUTCOMES:
Incidence of surgical site infection (SSI) at site of stoma closure | At seven days and 31 days after stoma closure
  The presence or not of surgical site infection (SSI) at site of stoma closure, evaluated at 7 and at 31 days after stoma closure according to the Center for Disease Control definition. Specialized nurses will record pictures of the stoma site for blinded evaluation by an investigator. In case of occurrence, SSI will be treated according to institutional guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Buchs, MD, PD, Study Director — University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meyer J, Delaune V, Abbassi Z, Douissard J, Toso C, Ris F, Buchs N. PROphylactic MESH (PROMESH) for stoma closure: does it reduce the incidence of incisional hernia? Protocol for a triple-blinded randomised controlled trial. BMJ Open. 2021 Dec 14;11(12):e053751. doi: 10.1136/bmjopen-2021-053751. PMID 34907065